CLINICAL TRIAL: NCT05155475
Title: Endoscopic Ultrasound Evaluation of the Common Bile Duct in Patients With Obstructive Jaundice Due to Bilio-pancreatic Malignancies: a Multicenter Prospective Study (ECCO Trial)
Brief Title: Endoscopic Ultrasound Evaluation of the Common Bile Duct in Patients With Obstructive Jaundice Due to Bilio-pancreatic Malignancies (ECCO Trial)
Acronym: ECCO
Status: Completed | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03461-54
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Obstructive Jaundice; Bilio-pancreatic Tumor
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with jaundice
  Interventions: Procedure: Ultrasound endoscopy

INTERVENTIONS:
Procedure: Ultrasound endoscopy — After identification of the lesion, the common bile duct will be identified and followed by the point of dilation due to the compression of the known lesion up to the hilum of the liver

SUMMARY:
To assess the size of the common bile duct in a large cohort of patients with jaundice following a malignant tumor of the head of the pancreas or the distal bile duct receiving a diagnostic EA for biopsy and / or for evaluation of tissue resectability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with jaundice and an injury to the head of the pancreas recommended for EUS-guided tissue acquisition or staging
* Patients with jaundice and distal CBD lesion suggestive of cholangiocarcinoma or Vater's ampulla carcinoma recommended for EUS-guided tissue acquisition or staging
* Serum bilirubin level ≥ 3 mg / dl
* Age ≥ 18 years old
* Subject affiliated or beneficiary of a social security scheme.
* Subject having been informed of this study and having given his no objection

Exclusion Criteria:

* Presence of altered anatomy due to previous gastric surgery (Billroth II or Roux-en-Y anastomosis)
* Sphincterotomy performed previously, plastic biliary stent or metal stent placement
* Percutaneous drainage of the bile ducts performed previously
* Pregnant, breastfeeding or parturient woman
* Protected patients: Adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision; hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old, with jaundice
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of the common bile duct size | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Jean Mermoz, Lyon, France